CLINICAL TRIAL: NCT00681876
Title: Phase II Study of Avastin Plus Erbitux Plus Irinotecan as 2nd Line Treatment of Locally Advanced or Metastatic Colorectal Cancer in Patients Achieving Disease Progression as Best Response After 1st Line Treatment With FOLFIRI+Avastin or XELIRI+Avastin
Brief Title: Phase II Study of Avastin + Erbitux + Irinotecan as 2nd Line Treatment of Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/05.32
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Colorectal Cancer
Keywords: Metastatic colorectal cancer; Second line; Irinotecan; Erbitux (Cetuximab); Avastin (Bevacizumab)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Irinotecan+Avastin+Erbitux
  Interventions: Drug: Irinotecan; Drug: Avastin; Drug: Erbitux

INTERVENTIONS:
Drug: Irinotecan — Irinotecan (IV) 150 mg/m2 on day 1 every two weeks until progression
  Other Names: CPT-11; Campto
Drug: Avastin — Avastin (IV) 10 mgr/Kgr on day 1 every 2 weeks until progression
  Other Names: Bevacizumab
Drug: Erbitux — Erbitux (IV)500 mg/m2 on day 1 every two weeks until progression
  Other Names: Cetuximab

SUMMARY:
This phase II study will evaluate the efficacy of the combination of two monoclonal antibodies (Avastin + Erbitux) with irinotecan, in patients with colorectal cancer progressed after 1st line treatment with FOLFIRI Avastin or XELIRI Avastin.

DETAILED DESCRIPTION:
Treating patients with primary resistance to the most active multi-agent combination remains a challenging clinical problem. The reported data demonstrated that addition of ERBITUX may reverse IRINOTECAN resistance. Further data support the feasibility of the combination of two monoclonal antibodies (AVASTIN+ERBITUX) with IRINOTECAN with better responses compared to historical controls (ERBITUX±IRINOTECAN). As such, a phase II study was designed to evaluate the efficacy of the combination of AVASTIN plus ERBITUX plus IRINOTECAN as second line treatment in patients progressing while on treatment with FOLFIRI AVASTIN or XELIRI AVASTIN

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic colorectal cancer.
* Measurable or evaluable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* ECOG performance status ≤ 2
* Age 18 - 72 years
* Patients with de novo refractory disease (progression of disease as best response at 1st line therapy with FOLFOX/Avastin)
* Adequate liver (Bilirubin ≤ 1.5 UNL, SGOT/SGPT ≤ 4 UNL, ALP ≤ 2.5 UNL),renal (Creatinine ≤ 1.5 UNL) and bone marrow (ANC ≥ 1,500/mm3, PLT ≥100,000/mm3) function
* Patients must be able to understand the nature of this study
* Written informed consent

Exclusion Criteria:

* History of serious cardiac disease (unstable angina, congestive heart failure, uncontrolled cardiac arrhythmias).
* History of myocardial infarction or stroke within 6 months.
* Clinically significant peripheral vascular disease.
* History of abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 28 days prior to Day 0.
* Presence of central nervous system or brain mets.
* Evidence of bleeding diathesis or coagulopathy.
* Patients with known hypersensitive reaction to cetuximab
* Blood pressure > 150/100 mmHg.
* Pregnant or lactating woman.
* Life expectancy < 3 months.
* Previous radiotherapy within the last 4 weeks or > 25% of bone marrow.
* Metastatic infiltration of the liver >50%.
* Patients with chronic diarrhea (at least for 3 months) or partial bowel obstruction or total colectomy.
* Active infection requiring antibiotics on Day 1.
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer.
* Psychiatric illness or social situation that would preclude study compliance.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Time To Progression | 1 year

SECONDARY OUTCOMES:
Objective Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)
Toxicity profile | Toxicity assessment on each chemotherapy cycle
Quality of life, Symptoms improvement | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: John Souglakos, MD, Principal Investigator — University Hospital of Crete
Locations (8):
- Greece (8):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - 401 Military Hospital of Athens, Athens
  - : "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - Air Forces Military Hospital of Athens, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - State General Hospital of Larissa, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki